CLINICAL TRIAL: NCT06032364
Title: Stone Disease of the Urinary Tract in Children: Clinical Presentation, Diagnostic Methods, Therapeutic Management, Evolution and Prognosis
Brief Title: Stone Disease of the Urinary Tract in Children
Acronym: Ped-Urolithia
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9020
Record Dates: First submitted 2023-08-31; First posted 2023-09-13 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Urinary Lithiasis
Keywords: Urinary Lithiasis; Stone disease; Urolithiasis; Urinary Calculi
MeSH Terms: conditions — Urolithiasis; Urinary Calculi

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of stone disease of the urinary tract in children is increasingly increasing with a remarkable economic impact for its management.

This incidence is variable according to race, geographic region, socio-economic status and dietary habits.

Oxalo-calcium stones are the most common but the biochemical nature of urinary stones varies depending on the region where those of a phosphatic nature are characterized by a higher incidence in Europe.

The diagnosis is confirmed by imaging. The unprepared abdomen (ASP) has low diagnostic accuracy. The scanner is the reference tool but remains an irradiating examination.

Risk factors for disease recurrence include primarily the presence of an underlying urinary metabolic abnormality and young age. Urinary metabolic abnormalities vary from one study to another.

The understanding of lithogenesis, its evaluation as well as the therapeutic options is essential for adequate and adapted management in the pediatric population.

ELIGIBILITY:
Inclusion criteria:

* Patients aged less than 18 years.
* Both sexes.
* Subjects presenting with lithiasis of the urinary tree in one of the two departments concerned between 01/01/2010 and 12/31/2022
* Subject not opposing, after information, the reuse of their data for the purposes of this research.
* Holders of parental authority who do not object, after being informed, to the reuse of their child's data for the purposes of this research.

Exclusion criteria:

* Subject or holder of parental authority having expressed opposition to participating in the study.
* Non-usable patient files: insufficient data.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged less than 18 years presenting with lithiasis of the urinary tree in one of the two departments concerned between 01/01/2010 and 12/31/2022
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-06-23 (Estimated); Study Completion 2025-06-23 (Estimated)

PRIMARY OUTCOMES:
Study of the modalities of the therapeutic management of children with urinary stones, retrospective description of the evolutionary aspects and the risk factors associated with recurrence. | Files analysed retrospectively from January 01, 2010 to December 31, 2022 will be examined
  This study is retrospective on already existing data

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pédiatrie 1 - CHU de Strasbourg - France, Strasbourg, France